CLINICAL TRIAL: NCT06643104
Title: Assessment of Adolescent Idiopathic Scoliosis Based on 3D Imaging With Depth Cameras: A Comparative Study of Back Height Difference and Angle of Trunk Rotation
Brief Title: 3D Imaging Assessment of Scoliosis: Back Height Difference vs. Trunk Rotation Angle
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KL-215-01-2
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BHD
  Interventions: Procedure: Tuina

INTERVENTIONS:
Procedure: Tuina — X-ray mapping guides three days of tailored exercises, including 3D therapy, breathing techniques, and spinal manipulation.
  Other Names: Tuina, sports gymnastics

SUMMARY:
This study focuses on adolescents with idiopathic scoliosis, employing 3D imaging technology with depth cameras to measure back height difference (BHD) and angle of trunk rotation (ATR) before and after conventional treatments such as massage, exercise therapy, and bracing. Statistical analyses are conducted to verify the correlation between BHD and ATR and to assess the sensitivity of BHD in evaluating short-term treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

(1) Adolescents aged 10-18 years, diagnosed with adolescent idiopathic scoliosis (AIS) with a Cobb angle ≥10°; (2) No history of spinal surgery or other corrective treatments; (3) Able to undergo short-term inpatient treatment (5 days) and comply with study procedures.

Exclusion Criteria:

(1) Patients with congenital, neuromuscular, or other secondary scoliosis; (2) Presence of major comorbidities affecting spinal structure or muscle tone (e.g., spinal cord injury, muscular dystrophy); (3) Patients unable to complete standardized assessment procedures.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study focuses on adolescents aged 10-18 diagnosed with adolescent idiopathic scoliosis, defined by a Cobb angle of ≥10°.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Back height difference | Day 1 of Admission and Day 5 of Admission
  Using depth cameras to acquire back data, point cloud processing algorithms analyze the information. The height difference between the highest point on the convex side and the corresponding point on the concave side is measured, with three repetitions taken to calculate the average value.

SECONDARY OUTCOMES:
Angle of trunk rotation | Day 1 of Admission and Day 5 of Admission
  A scoliometer is used to measure the patient's angle of trunk rotation (ATR). Measurements are repeated three times, and the average value is taken.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No